CLINICAL TRIAL: NCT06529471
Title: The Effect of Massage Applied After Open Cardiovascular Surgery on Patients' Pain, Sleep Quality and Serum Cortisol Level
Brief Title: Effect of Massage After CABG on Pain, Sleep Quality and Serum Cortisol Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, YASEMİN ÖZHANLI, Assist Prof, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/11.26; Kocaeli University (Other: Scientific Research Projects Coordination Unit)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Nursing Care; Massage; Pain; Cortisol
Keywords: massage; pain; nursing care; sleep; cortisol
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study was conducted experimentally with a pre-test and post-test control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blinding was used in the study. For this purpose, the participants were not specified in which group they belonged to the research. Therefore, a separate informed consent form was prepared for each group. In order to avoid bias in the analysis of the research data, statistician blinding was also applied.
  While coding the research data, the research groups were coded as A and B, and the statistician was prevented from knowing which letter represented which group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group receiving massage (Experimental): In Postoperative 0, before the massage, the patient's sleep duration (with the Richard-Campbell Sleep Scale and smart watch) and cortisol level are measured (first test). In Postoperative 1, a back massage is applied three times (10:00-14:00-20:00). In Postoperative 2, sleep duration (with the Richard-Campbell Sleep Scale and smart watch) and cortisol level are measured (last test).
  Interventions: Other: Massage group
- Standard care group (No Intervention): The patients in this group are given routine care practices of the clinic. Sleep and cortisol measurements are made in parallel with the experimental group.

INTERVENTIONS:
Other: Massage group — The patient in the massage group will be visited by the practitioner 3 times at 10:00-14:00-20:00 on the first day after surgery and a back massage will be applied. The patient in the massage group will be placed in an orthopnea position during the application. The massage procedure lasts an average of 30 minutes and is applied to the cervical 3 and thoracic 12 vertebrae.
  Arms: Group receiving massage

SUMMARY:
The patient in the surgical treatment and care process has difficulty in meeting the need for sleep in the hospital, and accordingly, their habits, attitudes and behaviors regarding sleep and rest change. Studies have shown that hospitalized patients experience sleep deprivatio.The decrease in sleep duration and quality is an important component affecting recovery after surgery. Studies have reported that massage reduces physical and emotional stress and increases sleep quality, while back massage reduces pain, anxiety and sleep disorders.

It has been reported that back massage reduces cortisol levels and blood pressure, slows heart rate and improves sleep quality (Pınar and Afşar 2015). This study was planned as a case-control study to evaluate the effect of massage therapy applied after open cardiovascular surgery on patients' pain, sleep quality and serum cortisol levels. It is thought that the study will create literature information on the sleep quality, pain and serum cortisol levels of patients after open heart surgery.

DETAILED DESCRIPTION:
Surgery is seen as an unexpected and negative experience in the lives of patients and their relatives. During the surgical procedure, the differences in the environment and lifestyle of patients, pain, changes in the body, the possibility of individual respect or disruption of body integrity may cause them to experience anxiety and fear. Patients in the treatment and care process have difficulty meeting their sleep needs in the hospital, and their habits, attitudes and behaviors regarding sleep and rest change accordingly.Studies have shown that hospitalized patients experience sleep deprivation. Different definitions of sleep have been made; however, according to the most common definition, sleep is a state of unconsciousness during the resting of the brain and from which the person can be awakened by external stimuli. Sleep, which has an important place in physical and mental health, has different aspects such as total duration, latency, regularity and quality. Sleep quality includes the quantitative (sleep latency, sleep duration, and number of awakenings per night) and qualitative (depth and restfulness of sleep) aspects of sleep. An average of 7-8 hours of sleep is needed daily and varies according to individual characteristics such as age, gender, nutrition, activity, health status, and physical environment, and accordingly, sleep quality can be affected both quantitatively and qualitatively. In the literature, it is reported that the sleep processes of hospitalized patients are negatively affected; this symptom is seen in 48-90% of patients in the postoperative period; and the cause of sleep problems is often pain. Surgical interventions affect the physiological and psychological health of patients and cause patients to experience great anxiety and fear about their lives and future. In addition, it is reported that general anesthetic drugs disrupt the sleep/wake cycle and other circadian rhythms such as body temperature and melatonin secretion. It is stated that sleep quality is low due to reasons such as postoperative pain, anxiety about the disease and positional restrictions after the intervention. Short and poor sleep duration reduces uninterrupted sleep and disrupts the 24-hour circadian rhythm and normal sleep pattern. In this sense, poor sleep quality can cause multi-system effects such as increased proinflammatory cytokines, blood pressure changes, increased risk of heart attack, hormonal stress response, glucose intolerance and suppression of the immune system. Therefore, the need for adequate sleep should be taken into account in both preoperative and postoperative care of surgical patients. Decreased sleep duration and quality is an important component affecting postoperative recovery. Because when combined with surgical stress, it can lead to increased catabolic activity and tissue destruction as well as decreased anabolic activity, which in turn affects postoperative recovery. Indeed, animal models have shown that sleep deprivation leads to depletion of glycogen stores and increases oxidative stress and free radical production, as well as the production of proinflammatory cytokines, all of which contribute to poor postoperative recovery. In a study conducted with patients in intensive care, it was reported that on average half of the patients had sleep problems and these problems continued after discharge, and that sleep problems in these clinics were pain, ventilation modes, and medications. In the study conducted by Sivas et al., it was stated that there was a significant relationship between pain, sleep disturbance, and quality of life. It was also determined that postoperative sleep quality was poor in patients who underwent cardiothoracic surgery and this situation lasted for more than 6 months. It is stated that patients in surgical clinics have low sleep quality due to reasons such as pain, anxiety related to the disease, encountering unknowns after surgery, and positional restrictions. Determining and eliminating the factors affecting the patient's sleep needs, ensuring and maintaining a normal sleep process are among the independent nursing roles. The stress response shows its effects by affecting vital organs and systems such as the central nervous, circulatory, gastrointestinal and immune systems, mainly through the autonomic nervous system and the hypothalamic-pituitary-adrenal (HPA) axis. Stress and the stress response can cause various clinically negative health outcomes (coronary artery disease, arrhythmia, memory problems, etc.). Numerous strategies have been developed and studied to alleviate the potential negative health effects of stress through effective management of stress with cognitive perceptual methods such as meditation, mindfulness and massage In addition to medical practices, nurses also use complementary practices to overcome symptoms such as insomnia, fatigue and pain. One of these practices, massage, is a simple, applicable, non-invasive method used to provide relaxation. The palpation of soft tissues and muscles provides both physical and mental relaxation for the person. In addition, massage is a therapeutic method that provides energy transmission between the nurse and the patient. Studies have reported that massage reduces physical and emotional stress and increases sleep quality, while back massage reduces pain, anxiety and sleep disorders. It has been reported that back massage reduces cortisol levels and blood pressure, slows down heart rate and increases sleep quality. This study was planned as a case-control study to evaluate the effect of massage applied after open heart surgery on pain, sleep quality and serum cortisol levels of patients. It is thought that the study will create literature information on the sleep quality, pain and serum cortisol levels of patients applied after open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planning for elective open heart surgery
* Being conscious
* Being extubated

Exclusion Criteria:

* Those who underwent minimally invasive cardiac surgery,
* Those who did not use an extracorporeal circulation machine
* Those who have an infectious disease such as varicella zoster on the back, or a structural disease such as scoliosis,
* Those who have another surgical procedure performed simultaneously on the back,
* Those who have no limb loss

Ages: 40 Years to 71 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | Before the recruit pre-test (RCSQ- survey scale) will be applied. A post-test (RCSQ survey scale) will be administered again two days after the intervention.]
  Richard-Campbell Sleep Scale: RCSQ is a 6-item scale that evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time it takes to stay awake when you wake up, the quality of sleep, and the noise level in the environment. Each item is evaluated on a chart from 0 to 100 using the visual analog scale technique. A score between "0-25" from the scale indicates very poor sleep, and a score between "76-100" indicates very good sleep. The total score of the scale is evaluated over 5 items, and the 6th item, which evaluates the noise level in the environment, is excluded from the total score evaluation. As the score of the scale increases, the sleep quality of the patients also increases.
Postoperative Pain Intensity (Numeric Rating Scale) | Measured before each session and 10 minutes after each session, as well as on postoperative days 1 and 2.
  Postoperative pain intensity will be assessed using the 0-10 Numeric Rating Scale, where 0 indicates "no pain" and 10 indicates "worst possible pain." Pain will be measured at standardized time points for all participants. In the intervention group, pain will be assessed immediately before each massage session and 10 minutes after each session. In the control group, pain assessments will follow the same schedule corresponding to routine care time points. Higher scores indicate greater pain severity.

SECONDARY OUTCOMES:
Secondary Outcome Measure | Before the recruit pre-test (serum cortisol-blood test) will be applied. A post-test (serum cortisol-blood test) will be administered two days after the intervention.]
  Serum Cortisol Level Analysis: Blood samples will be placed in tubes containing separator gel (SST-yellow tube) and serum cortisol levels will be analyzed in the relevant laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No